CLINICAL TRIAL: NCT00691613
Title: Infusion of a Single Dose of Erythropoietin to Prevent Injury in an Ischemia Reperfusion Forearm Model - A Randomised Cross-over Study to Evaluate if Infusion of a Single Dose of EPO Protects Against Ischemia-reperfusion Injury in Man
Brief Title: Infusion of a Single Dose of Erythropoietin to Prevent Injury in an Ischemia Reperfusion Forearm Model
Acronym: IPIIR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Medical Center Groningen (Other)
Collaborators: Radboud University Medical Center (Other)
Responsible Party: Prof. dr. W.H. van Gilst, University Medical Centre Groningen, Dept. of Cardiology
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: WTR-ECG-3; EudraCT 2007-001089-33
Record Dates: First submitted 2008-06-03; First posted 2008-06-05 (Estimated); Last update posted 2010-03-12 (Estimated); Status verified 2010-03

CONDITIONS: Ischemia-Reperfusion Injury; Myocardial Infarction
Keywords: Apoptosis; Annexin; Hypoxia; Ischemia-Reperfusion Injury
MeSH Terms: conditions — Reperfusion Injury; Myocardial Infarction; Hypoxia | interventions — Epoetin Alfa; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): EPO
  Interventions: Drug: Epoetin alpha
- 2 (Placebo Comparator): NaCl
  Interventions: Drug: NaCl

INTERVENTIONS:
Drug: Epoetin alpha — The dosage (60.000 I/U Epoetin alpha) will be diluted in 10 ml of 0.9% sodium chloride solution and injected in a single dose intravenously in the dominant forearm (the non-dominant forearm will be used as ischemic model).
  Other Names: Eprex
  Arms: 1
Drug: NaCl — 0.9% sodium chloride solution as placebo dosage is 10 ml, which will be administered in the same manner as the interventional medicinal product.
  Other Names: Sodiumchloride, saline
  Arms: 2

SUMMARY:
Rationale:

The investigators hypothesize that EPO protects against apoptosis after acute ischemia in man and that it is detectable using the annexin-A5 model.

Objective:

Does infusion of a single dose of Epoetin Alfa, a short-acting EPO, protect against apoptosis in man after acute ischemia?

Study design:

A double blinded randomised cross-over study.

Study population:

12 Healthy male volunteers, between 18 and 40 years old.

Intervention:

All 12 volunteers will receive a single dose of EPO and placebo in a randomized order. A six week wash-out period is obtained in order to avoid interference of both treatments.

Main study parameters/endpoints:

The percentage of difference between radioactivity (quantified as counts per pixel) of the experimental and control thenar muscle at one and four hours after reperfusion.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers between 18 and 40 years of age
* male
* Volunteers are not allowed smoking 24 hours before the start of the experiment

Exclusion Criteria:

* Female
* Hypertension (SBP >140 mmHg, DBP >90 mmHg)
* Diabetes Mellitus (DM) (fasting glc >6.9 mmol/l, glc >11.0 mmol/l)
* Hypercholesterolemia
* Renal dysfunction (eGFR < 60 ml/min, calculated using MDRD formula)
* Any known hypersensitivity/allergic reaction to one of the constituents of Epoetin Alfa
* A history of use of any form of EPO
* Any current medication use
* Cardiovascular disease in medical history
* Smoking less than 24 hours prior to Epoetin alpha infusion
* Participation in research in the last 5 years in which any form of radioactivity was used
* No participation in any research trial in the last 30 days or 5 times the half-life of the used substance

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2010-07; Primary Completion 2011-10 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
The percentage of difference between radioactivity (quantified as counts per pixel) of the predefined area of interest of the experimental and control thenar muscle at one and four hours after reperfusion. | 4 hours

SECONDARY OUTCOMES:
DNA polymorphisms affecting HO-1 and AMP-deaminase activity is assessed by DNA analysis. | 4 hours
The effect of EPO treatment on heme oxygenase activity as measured in blood and as CO concentration in exhaled air. | 4 hours
Maximal voluntary contraction and duration of the exercise during ischemia. | 10 minutes

CONTACTS AND LOCATIONS:
Overall Officials: W. H. van Gilst, Prof, PhD, Study Chair — University Medical Center Groningen; P. Smits, Prof, MD, PhD, Study Chair — University Medical Centre Nijmegen; W. T. Ruifrok, MD, Principal Investigator — University Medical Center Groningen; G. A. Rongen, MD, PhD, Study Director — University Medical Centre Nijmegen; D.J. van Veldhuisen, Prof, MD, PhD, Study Director — University Medical Center Groningen; W. Oyen, Prof, MD, PhD, Principal Investigator — University Medical Centre Nijmegen; R. A. de Boer, MD, PhD, Principal Investigator — University Medical Center Groningen; P.P. van Geel, MD, PhD, Principal Investigator — University Medical Center Groningen; R. A. Tio, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- Clinical Research Centre Nijmegen, Nijmegen, Gelderland, Netherlands

REFERENCES:
- See also: Webpage of the University Medical Centre Nijmegen — http://www.umcn.nl